CLINICAL TRIAL: NCT01983657
Title: Study of Subcutaneous Injection of Low-dose Recombinant Granulocyte Macrophage-Colony Stimulating Factor (rhGM-CSF) +/- Whole Lung Lavage(WLL) in Pulmonary Alveolar Proteinosis.
Brief Title: Study of Subcutaneous Injection of Low-dose rhGM-CSF +/- WLL in PAP.
Acronym: PAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Huiping Li, Professor,Chief of Dept. of Respiratory Medicine, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120401
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Pulmonary Alveolar Proteinosis
Keywords: Pulmonary; Pulmonary Alveolar Proteinosis; PAP
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis | interventions — regramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- D1 (Experimental): Patients diagnosed with PAP will be received rhGM-CSF 1.25 ug/kg/d subcutaneously for 1 month, before evaluation on the 30th day (±3 day).
  If the treatment is effective, participants may be entered into low-dose group(D1)(rhGM-CSF administration 1.25 ug/kg/d, qd, sc, for 2 months，then rhGM-CSF administration 1.25 ug/kg/d, qod, sc, for 3 months), when the chest CT absorption≥25% , and /or the PaO2 elevated by 5 mm Hg.
  Interventions: Drug: rhGM-CSF
- D2 (Experimental): Patients diagnosed with PAP will be received rhGM-CSF 1.25 ug/kg/d subcutaneously for 1 month, before evaluation on the 30th day (±3 day).
  When the treatment is ineffective, and anti-GM-CSF antibody titers level ≥1:1000，the dose will be increased to 2.5 ug/kg/d. After 2 months, if the clinical response was optimal, that dose is continued for 3 months, and defined as group 2(D2).
  Interventions: Drug: rhGM-CSF
- D3 (Experimental): Patients diagnosed with PAP will be received rhGM-CSF 1.25 ug/kg/d subcutaneously for 1 month, before evaluation on the 30th day (±3 day).
  When the treatment is ineffective, and anti-GM-CSF antibody titers level ≥1:1000，the dose will be increased to 2.5 ug/kg/d. After 2 months, if the clinical response was not optimal, the patients will receive whole lung lavage(WLL), who are defined as group 3(D3).
  Interventions: Drug: rhGM-CSF
- D4 (Active Comparator): Patients diagnosed with PAP will be received rhGM-CSF 1.25 ug/kg/d subcutaneously for 1 month, before evaluation on the 30th day (±3 day).
  When the treatment is ineffective, and anti-GM-CSF antibody titers level <1:1000，the patients will receive whole lung lavage(WLL), then give rhGM-CSF administration (1.25 ug/kg/d) for 3 months, which belong to group4(D4).
  Interventions: Drug: rhGM-CSF; Procedure: Whole Lung Lavage(WLL)

INTERVENTIONS:
Drug: rhGM-CSF — GM-CSF will be given subcutaneously according to the rule in different groups.
  Other Names: TOPLEUCON; GM-CSF; Recombinant Granulocyte Macrophage-Colony Stimulating Factor; Granulocyte Macrophage-Colony Stimulating Factor
Procedure: Whole Lung Lavage(WLL) — using double lumen endotracheal tube (DLT) to selectively lavage one lung
  Other Names: Whole Lung Lavage; WLL
  Arms: D4

SUMMARY:
The purpose of this study is to establish an efficient and economic treatment scheme by evaluation of the safety and efficacy of subcutaneous injection of low-dose rhGM-CSF, or of similar injection after whole lung lavage , in patients with PAP.

DETAILED DESCRIPTION:
The purpose of this study is to establish an efficient and economic treatment scheme by evaluation of the safety and efficacy of subcutaneous injection of low-dose rhGM-CSF, or of similar injection after whole lung lavage , in patients with PAP. During the observation, study visits will occur at the end of each month. During the 1-year follow-up period which is lasting 6 months after the treatment, all participants will be required to check the various efficacy indicators.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed PAP patients
* Aged 17-80
* Signed informed consent

Exclusion Criteria:

* Secondary PAP
* Received whole lung lavage therapy within 4 weeks before enrollment
* Received previous GM-CSF therapy within 6 months before enrollment
* WBC≥12,000/ul
* fever≥38℃
* Severe edema, severe liver, kidney, lung and cardiovascular disease.
* Pregnant，planning to get pregnant or nursing
* Inability to express the subjective discomfort
* Serious drug allergy history, E.coli preparation or rhGM-CSF serious allergy history

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Improvements in double pulmonary diffuse lesions （Chest CT score ） | 6 months

SECONDARY OUTCOMES:
Clinical symptoms observation: shod of breath, cough (according to each score standard） | 6 months
Granulocyte Macrophage Colony Stimulating Factor(GM-CSF) Antibody titer change | 6 months
Improvements in pulmonary function | 6 months
  Pulmonary function tests include residual volume/total lung capacity(RV/TLC), forced vital capacity(FVC), forced expiratory volume in one second/forced vital capacity(FEV1/FVC), diffusing capacity of carbon monoxide(DLCO).
Improvements in arterial blood gas, including alveolar-arterial oxygen difference(A-aDO2), partial pressure of oxygen(PaO2), partial pressure of carbon dioxide in artery(PaCO2), arterial oxygen saturation(SaO2). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Huiping Li, Dr, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

REFERENCES:
- [Derived] Zhang F, Weng D, Su Y, Yin C, Shen L, Zhang Y, Zhou Y, Li Q, Hu Y, Li H. Therapeutic effect of subcutaneous injection of low dose recombinant human granulocyte-macrophage colony-stimulating factor on pulmonary alveolar proteinosis. Respir Res. 2020 Jan 2;21(1):1. doi: 10.1186/s12931-019-1261-1. PMID 31898493